CLINICAL TRIAL: NCT02993978
Title: Design and Evaluation of Care Environment and Technology at Pediatric Radiotherapy
Acronym: DUMBO
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-113-31M
Record Dates: First submitted 2016-11-21; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-11

CONDITIONS: Pediatric ALL; Radiotherapy Side Effect
Keywords: Pediatric radiotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Pediatric patients and their parents who were treated with radiotherapy during baseline period and enrolled in the study. Recruitment to the Control Group took Place during one year.
- Case group: Pediatric patients and their parents who were treated with radiotherapy during case period and enrolled in the study. Recruitment to the case group took place during one year after introduction of new methods and equipment in the in the clinic..

SUMMARY:
The purpose of the study is to evaluate the effect of changes in the care environment in pediatric radiotherapy. The definitions of the changes is a part of the study, and is constructed in collaboration with the institute of design at Umeå University. The implementation is however not part of the study, but done as part of Clinical routine.

The study consist of two parts, where the first 1.5 years are a Control phase where the changes are designed and also function as a baseline period. The following 1.5 years are the case period where the Changes that are accepted for Clinical implementation are implemented.

The impact of the changes are evaluated using surveys and interviews of both parents and children

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effect of changes in the care environment in pediatric radiotherapy. The definitions of the changes is a part of the study, and is constructed in collaboration with the institute of design at Umeå University. The implementation is however not part of the study, but done as part of Clinical routine.

The study consist of two parts, where the first 1.5 years are a Control phase where the changes are designed and also function as a baseline period. The following 1.5 years are the case period where the Changes that are accepted for Clinical implementation are implemented.

The impact of the changes are evaluated using surveys and interviews of both parents and children. Interviews of the personnel regarding their experiences of the study and the changes is performed after the finalization of the case period.

ELIGIBILITY:
Inclusion Criteria:

* Radiotherapy treatment

Exclusion Criteria:

-

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients treated with radiotherapy at the study centres were candidates for the study.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Parents anxiety during treatment period | 1 day
  VAS-anxiety scoring in connection to therapy
Childrens anxiety during treatment period | 1 day
  FAS-evaluation
Parents quality of Life during treatment period | 1 day
  PedsQL survey
Parents view of the care and care environment | After treatment period (within 2 months after last treatment)
  Semi structured interview
Childrens reflections regarding the treatment period | After treatment period (within 2 months after last treatment)
  Semi structured interview

SECONDARY OUTCOMES:
Use of sedative treatment in connection to radiotherapy | up to 2 months
  The use of sedative treatments were recorded for each fraction
Experiences of the personnel | After the case period (within 1 year)
  Interviews

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Engvall G, Angstrom-Brannstrom C, Mullaney T, Nilsson K, Wickart-Johansson G, Svard AM, Nyholm T, Lindh J, Lindh V. It Is Tough and Tiring but It Works--Children's Experiences of Undergoing Radiotherapy. PLoS One. 2016 Apr 7;11(4):e0153029. doi: 10.1371/journal.pone.0153029. eCollection 2016. PMID 27055258
- [Result] Angstrom-Brannstrom C, Engvall G, Mullaney T, Nilsson K, Wickart-Johansson G, Svard AM, Nyholm T, Lindh J, Lindh V. Children Undergoing Radiotherapy: Swedish Parents' Experiences and Suggestions for Improvement. PLoS One. 2015 Oct 28;10(10):e0141086. doi: 10.1371/journal.pone.0141086. eCollection 2015. PMID 26509449
- [Derived] Engvall G, Lindh V, Mullaney T, Nyholm T, Lindh J, Angstrom-Brannstrom C. Children's experiences and responses towards an intervention for psychological preparation for radiotherapy. Radiat Oncol. 2018 Jan 22;13(1):9. doi: 10.1186/s13014-017-0942-5. PMID 29357940